CLINICAL TRIAL: NCT01838811
Title: Applying Speed of Processing Training (SPT) to Individuals With TBI
Brief Title: Applying Speed of Processing Training to Individuals With Traumatic Brain Injury
Acronym: SPTTBI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kessler Foundation (Other)
Responsible Party: Principal Investigator, Nancy Chiaravalloti, Director, Neuropsychology & Neuroscience Lab, Kessler Foundation
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: KF 30.01
Record Dates: First submitted 2012-05-11; First posted 2013-04-24 (Estimated); Last update posted 2015-04-03 (Estimated); Status verified 2015-04

CONDITIONS: Traumatic Brain Injury
Keywords: Processing Speed; Intervention; Traumatic Brain Injury; Cognition
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Speed of Process Training — SPT involves trainer-guided practice of computer-based exercises, including Target Detection (indicating presence or absence of targets, identifying targets, etc.) and Discrimination and Localization (performing same/ different discriminations of targets presented very quickly and followed by a masking pattern) 10, 19, 84. Display speed, ranging from 17 to 500 ms, is the primary manipulation during training, which increases task demands and thus demands on PS itself. These training tasks are tailored to each individual's ability by the trainer.

SUMMARY:
This pilot study will document the efficacy of a behavioral intervention for Processing Speed (PS) in Traumatic Brain Injury (TBI), Speed of Processing Training (SPT), which has been successful used in the aging population in several studies. This study will (1) apply a treatment protocol for PS impairments, well-validated in aging, to persons with TBI with impaired PS, and document its efficacy on standard neuropsychological (NP) tests (2) assess the effectiveness of the intervention utilizing global measures of daily life, including an objective measure (TIADL) (3) examine the long term impact of SPT. This study is unique in that it will be the first to evaluate the efficacy of a highly-manualized structured behavioral treatment for processing speed deficits in persons with TBI utilizing the optimal methodology for carrying out such studies, a randomized clinical trial. Given the prevalence of PS deficits in the TBI population and the significant impact such deficits have on everyday functioning, public safety, and overall quality of life, the identification of an effective intervention for PS deficits in TBI could have a profound impact on the population and society as a whole.

ELIGIBILITY:
Inclusion Criteria:

* fluent in English
* processing speed impairment (based on evaluation).

Exclusion Criteria:

* currently taking steroids and /or benzodiazepines
* prior stroke or neurological disease
* history of significant psychiatric illness (for example, bipolar disorder, schizophrenia, or psychosis) or a current diagnosis of Major Depressive Disorder, Schizophrenia, Bipolar Disorder I or II.
* significant alcohol or drug abuse history

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2011-11; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Processing Speed Performance | week 6 and week 12
  Neuropsychological tests which measure processing speed will be used to determine whether there has been a change in performance.

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Chiaravalloti, Ph.D., Principal Investigator — Kessler Foundation
Locations (1):
- Kessler Foundation, West Orange, New Jersey, United States